CLINICAL TRIAL: NCT03583164
Title: Phase IIb Study of F901318 as Treatment of Invasive Fungal Infections Due to Lomentospora Prolificans, Scedosporium Spp., Aspergillus Spp., and Other Resistant Fungi in Patients Lacking Suitable Alternative Treatment Options
Brief Title: Evaluate F901318 (Olorofim) Treatment of Invasive Fungal Infections in Participants Lacking Treatment Options
Acronym: FORMULA-OLS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F901318/0032
Record Dates: First submitted 2018-05-17; First posted 2018-07-11 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Invasive Fungal Infections
Keywords: Anti fungal; Invasive aspergillosis; Rare moulds; Coccidioidomycosis
MeSH Terms: conditions — Invasive Fungal Infections; Coccidioidomycosis | interventions — olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olorofim (F901318) (Experimental): Olorofim (F901318) was given orally for up to 90 days in the Main Study Phase and could be continued for those participants entering the Extended Treatment Phase.
  Patients received fixed doses comprising of a 1-day loading dose of 150 mg of olorofim twice a day followed by a maintenance dose of 90 mg of olorofim twice a day.
  Up until Protocol Amendment 06, 58 patients received a weight-based olorofim dosing consisting of a 1-day loading dose of 4 mg/kg/day on Day 1, then a maintenance dose of 2.5 mg/kg/day (divided into 2 or 3 doses). The dose was then adjusted based on plasma levels of olorofim with the maximum total daily dose of 300 mg.
  Interventions: Drug: Olorofim

INTERVENTIONS:
Drug: Olorofim — 30mg oral tablets
  Other Names: F901318

SUMMARY:
A study to evaluate olorofim (F901318) for the treatment of invasive fungal infections in participants lacking suitable alternative treatment options.

DETAILED DESCRIPTION:
An open label, single arm Phase IIb study of olorofim (F901318) in participants with invasive fungal infections with limited treatment options. Participants received study treatment for up to 12 weeks in the main phase of the study. At the Investigator's request and after discussion with the medical monitor, open-label treatment with F901318 could be continued in patients judged by the Investigator to need therapy beyond 84 days and considered likely to continue to benefit from extended treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged at least 18 years, or male and female aged 16 years or 17 years and who weigh at least 40 kg whom have given informed consent
* Ability and willingness to comply with the protocol.
* Able to take oral medication
* Females must be non-lactating and at no risk of pregnancy
* Male with female partners of childbearing potential must either abstain from sexual intercourse or use a highly effective means of contraception
* Participants with invasive fungal disease
* Participants who have limited alternative treatment options

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Known history of allergy, hypersensitivity, or any serious reaction to any component of the study drug.
* Participants with chronic aspergillosis, aspergilloma or allergic bronchopulmonary aspergillosis.
* Human Immunodeficiency Virus (HIV) infection but not currently receiving antiretroviral therapy.
* Participants with a medical condition that may jeopardize adherence to the protocol or may cause unacceptable additional risk to the participant
* Previously enrolled participants or participants enrolled in any clinical trial within the last 30 days
* Participants receiving treatment limited to supportive care due to predicted short survival time.
* Prohibited concomitant medications.
* Any exclusion criteria required by local regulatory authorities.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chen, Principal Investigator — Westmead Hospital
Locations (82):
- United States (14):
  - Valley Fever Institute at Kern Medical Center, Bakersfield, California
  - UC Davis Medical Center, Sacramento, California
  - University of California San Diego Medical Center, San Diego, California
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Health System, Durham, North Carolina
  - UPMC, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Australia (6):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Peter MacCallum Centre-East Melbourne, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - UZ Leuven, Leuven, Waals-Brabant
  - Institut Jules Bordet, Brussels
  - Hôpital Erasme, Brussels
- Brazil (9):
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - HC - UFPR - Hospital de Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital da Universidade Federal de Santa Maria CEP/UFSM, Santa Maria, Rio Grande do Sul
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba
  - Santa Casa de Misericórdia de Passos, Passos
- Egypt (7):
  - Oncology Center, Mansoura University, Al Mansurah
  - Alexandria University Hospital, Alexandria
  - Cairo University Hospitals, Cairo
  - Ain Shams University Hospital, Cairo
  - Air Force Specialized Hospital, Cairo
  - National Cancer Institute, Cairo
  - Nasser Institute, Cairo
- France (4):
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble, Isere
  - Hôpital Necker - Enfants Malades, Paris, Paris
  - Hôpital Saint-Louis, Paris
- Germany (4):
  - Klinikum der Universitaet Muenchen Campus Grosshadern, Munich, Bavaria
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite-Campus Benjamin Franklin (CBF), Berlin
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (3):
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht, Utrecht
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Russia (4):
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - SBEIHPE "NWSMU n. a. I.I Mechnikov" of MoH and SD of RH, Saint Petersburg
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Thailand (2):
  - Siriraj Hospital, Bangkoknoi, Bangkok
  - King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok
- Turkey (Türkiye) (3):
  - Dicle University, Medical Faculty, Diyarbakır
  - Acibadem Atakent Hospital, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
- United Kingdom (3):
  - King's College Hospital, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Wythenshawe Hospital, Manchester, Wythenshawe
- Vietnam (4):
  - Bach Mai Hospital, Hanoi
  - National Lung Hospital, Hanoi
  - HCMC Hospital for Tropical Diseases, Ho Chi Minh City
  - Blood Transfusion Hematology Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results can be available to researchers after the primary publication of results for this study, after deidentification (text, tables, figures, appendices)
Supporting Information: Study Protocol, SAP
Time Frame: From 3 months after publication of the primary manuscript (no end date)
Access Criteria: Requests should be directed to F2G for review.

REFERENCES:
- [Derived] Maertens JA, Thompson GR 3rd, Spec A, Donovan FM, Hammond SP, Bruns AHW, Rahav G, Shoham S, Johnson R, Rijnders B, Schaenman J, Hoenigl M, Morrissey CO, Mehta SR, Heath CH, Koehler P, Paterson DL, Slavin MA, Fortun J, Nguyen MH, Patterson TF, Uspenskaya O, Van de Veerdonk FL, Verweij PE, Aoun M, Georgala A, Alexander BD, Chayakulkeeree M, Mehra V, Miceli MH, Sikka MK, Sole A, Walsh TJ, Aguado JM, Holland SM, Moussa M, Rautemaa-Richardson R, Bazaz R, Schwartz S, Walsh SR, Plate M, Yehudai-Ofir D, Bruggemann RJ, Cornely OA, Ostrosky-Zeichner L, Vazquez JA, White PL, Cornelissen K, Ross GG, Fitton L, Dane A, Zinzi D, Rex JH, Chen SC. Olorofim for the treatment of invasive fungal diseases in patients with few or no therapeutic options: a single-arm, open-label, phase 2b study. Lancet Infect Dis. 2025 Nov;25(11):1177-1188. doi: 10.1016/S1473-3099(25)00224-5. Epub 2025 Jun 18. PMID 40541222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study planned to enrol approximately 200 patients at approximately 100 centres globally over at least 60 months. The first patient was enrolled into the study on 06 June 2018 and the Last subject last visit date was 10 February 2023 (for the Extended Treatment Phase).
Groups:
- Olorofim (F901318): Open-label single-arm of F901318 (olorofim) as treatment of invasive fungal infections due to Lomentospora prolificans, Scedosporium spp., Aspergillus spp., and other resistant fungi which are susceptible to F901318 in patients with limited treatment options.
  Olorofim 30 mg tablets were given for up to 90 days in the Main Study Phase and could be continued for those entering the Extended Treatment Phase.
  Patients received a 1-day loading dose of 150 mg of olorofim twice a day followed by a maintenance dose of 90 mg of olorofim twice a day.
  Up until Protocol Amendment 06, 58 patients received a weight-based olorofim dosing consisting of a 1-day loading dose of 4 mg/kg/day on Day 1, then a maintenance dose of 2.5 mg/kg/day (divided into 2 or 3 doses). The dose was then adjusted based on plasma levels of olorofim with the maximum total daily dose of 300 mg.
Period: Overall Study
Arm/Group | Olorofim (F901318)
Started | 203
Completed | 126
Not Completed | 77
Not completed — Death in Main Phase | 35
Not completed — Lost to Follow up in Main Phase | 1
Not completed — Lost to follow up in Extended Phase | 3
Not completed — Clinically significant lab value in Main Phase | 2
Not completed — Clinically significant lab value in Extended Phase | 4
Not completed — Physician decision in Main Phase | 1
Not completed — Physician decision in Extended Phase | 2
Not completed — Death in Extended Phase | 13
Not completed — Intolerable adverse event in Main Phase | 3
Not completed — Intolerable adverse event in Extended Phase | 1
Not completed — Lack of compliance in Extended Phase | 2
Not completed — Treatment failure in Main Phase | 2
Not completed — Treatment failure in Extended Phase | 4
Not completed — Withdrawal of consent in Extended Phase | 2
Not completed — Other not specified reason in Main Phase | 2

BASELINE CHARACTERISTICS:
Groups:
- Olorofim (F901318): Open-label single-arm of Olorofim (F901318) as treatment of invasive fungal infections due to Lomentospora prolificans, Scedosporium spp., Aspergillus spp., and other resistant fungi which are susceptible to F901318 in patients with limited treatment options.
  Olorofim 30 mg tablets were given for up to 90 days in the Main Study Phase and could be continued for those entering the Extended Treatment Phase.
  Patients received fixed doses comprising of a 1-day loading dose of 150 mg of olorofim twice a day followed by a maintenance dose of 90 mg of olorofim twice a day.
  Up until Protocol Amendment 06, 58 patients received a weight-based olorofim dosing consisting of a 1-day loading dose of 4 mg/kg/day on Day 1, then a maintenance dose of 2.5 mg/kg/day (divided into 2 or 3 doses). The dose was then adjusted based on plasma levels of olorofim with the maximum total daily dose of 300 mg.
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 151
  >=65 years | 52
Age, Continuous [Median (Full Range); unit: years] | 56.57 [18.0 to 90.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 16
  White | 160
  More than one race | 2
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 96
  Egypt | 1
  United Kingdom | 3
  Thailand | 2
  Spain | 6
  Russia | 3
  Netherlands | 16
  Belgium | 45
  Israel | 8
  Australia | 18
  Germany | 5
Body Mass Index [Median (Full Range); unit: kg/m^2] | 22.954 [14.21 to 43.23]
Baseline Data Review Committee-Adjudicated Disease Category [Count of Participants; unit: Participants]
  Aspergillus - All | 101
  Lomentospora (Scedosporium) prolificans | 26
  Scedosporium spp. | 22
  Other Olorofim-susceptible fungi | 12
  Coccidioides | 41
  No DRC adjudicated baseline fungus | 1
Reason for Limited Treatment Options [Count of Participants; unit: Participants]
  Known/predicted resistance to all licensed agents | 42
  Failure of available therapy | 110
  Intolerance to available therapy | 29
  Inability to manage drug interactions | 7
  Inability to produce therapeutic drug levels | 2
  IV only option produced clinical response and standard to switch to oral azole | 10
  Other, received Medical Monitor approval | 2
  Missing | 1
Duration from Baseline Fungal Infection Start to First Treatment Administration [Median (Full Range); unit: Days] | 75.0 [1 to 3821]

OUTCOME MEASURES:

1. Primary Outcome: Data Review Committee (DRC) Adjudicated Overall Response at Day 42
Description: The primary efficacy variable was the DRC-adjudicated overall response at the Day 42 Study Visit, as determined by an independent DRC using a combination of clinical, mycological, and radiological results based on European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) criteria. For the primary statistical analysis of overall response rate, values were assigned to the DRC adjudicated overall response as follows: Success (Success-Complete, Success-Partial); Failure (Failure-Stable, Failure-Progression, Death, and participants for whom data at the Day 42 Study Visit could not be collected or participants who were considered not evaluable at the Day 42 Study Visit).
Time Frame: Day 42 in the Main Phase of study treatment
Population: The modified Intent to Treat (mITT) analysis set contains all participants in the ITT set who were assigned to a DRC-adjudicated disease category. The mITT population and subpopulations based on the DRC-adjudicated disease categories were used for the analysis of efficacy data.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Groups:
- Olorofim (F901318): Single arm open label olorofim treatment.
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 28.7 [22.6 to 35.5]

2. Secondary Outcome: DRC Adjudicated Overall Response at Day 42 for All Aspergillus
Description: The primary efficacy variable was the DRC-adjudicated overall response at the Day 42 Study Visit, as determined by an independent DRC using a combination of clinical, mycological, and radiological results based on EORTC/MSG criteria. This was also presented by each of the 5 major infections as adjudicated by the DRC at baseline. The Aspergillus- All category is a combination of participants with Aspergillus proven and Aspergillus probable (invasive aspergillosis lower respiratory tract disease) baseline disease category. Overall success is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT subpopulation contains all participants in the ITT set who had a DRC-adjudicated baseline infection of All Aspergillus.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 101
Response rate percentage | 34.7 [25.5 to 44.8]

3. Secondary Outcome: DRC Adjudicated Overall Response at Day 42 for Lomentospora Prolificans
Description: The primary efficacy variable was the DRC-adjudicated overall response at the Day 42 Study Visit, as determined by an independent Data Review Committee using a combination of clinical, mycological, and radiological results based on EORTC/MSG criteria. This was also presented by each of the 5 major infections as adjudicated by the DRC at baseline, this one is for participants with a proven infection due to Lomentospora prolificans. Success is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main Phase of study treatment Day 42 in the Main Phase of study treatment Day 42 in the Main Phase of study treatment Day 42 in the Main Phase of study treatment Day 42 in the Main Phase of study treatment
Population: The mITT subpopulation contains all participants in the ITT set who had a DRC-adjudicated baseline infection due to Lomentospora prolificans.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 26
Response rate percentage | 42.3 [23.4 to 63.1]

4. Secondary Outcome: DRC Adjudicated Overall Response at Day 42 for for Scedosporium Species
Description: The primary efficacy variable was the DRC-adjudicated overall response at the Day 42 Study Visit, as determined by an independent DRC using a combination of clinical, mycological, and radiological results based on EORTC/MSG criteria. This was also presented by each of the 5 major infections as adjudicated by the DRC at baseline, this one is for participants with a proven infection due to Scedosporium species. Success is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT subpopulation contains all participants in the ITT set who had a DRC-adjudicated baseline infection due to Scedosporium species.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 22
Response rate percentage | 36.4 [17.2 to 59.3]

5. Secondary Outcome: DRC Adjudicated Overall Response at Day 42 for Coccidioides Species
Description: The primary efficacy variable was the DRC-adjudicated overall response at the Day 42 Study Visit, as determined by an independent DRC using a combination of clinical, mycological, and radiological results based on EORTC/MSG criteria. This was also presented by each of the 5 major infections as adjudicated by the DRC at baseline, this one is for participants with proven infection due to Coccidioides species. Success is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT subpopulation contains all participants in the ITT set who had a DRC-adjudicated baseline infection due to Coccidioides species.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 41
Response rate percentage | 0.0 [0.0 to 8.6]

6. Secondary Outcome: DRC Adjudicated Overall Response at Day 42 for Other Olorofim Susceptible Fungi
Description: The primary efficacy variable was the DRC-adjudicated overall response at the Day 42 Study Visit, as determined by an independent DRC using a combination of clinical, mycological, and radiological results based on EORTC/MSG criteria. This was also presented by each of the 5 major infections as adjudicated by the DRC at baseline, this one is for participants with proven infection due to other olorofim susceptible fungi. Success is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT subpopulation contains all participants in the ITT set who had a DRC-adjudicated baseline infection due to other olorofim susceptible fungi.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 12
Response rate percentage | 33.3 [9.9 to 65.1]

7. Secondary Outcome: DRC Adjudicated Overall Response at Day 84
Description: DRC-adjudicated overall response at Day 84, as determined by an independent DRC using a combination of clinical, mycological, and radiological results based on the EORTC/MSG criteria. For the analysis of overall response rate, values were assigned to the DRC-adjudicated overall response as follows: Success (Success-Complete, Success-Partial); Failure (Failure-Stable, Failure-Progression, Death, and participants for whom data at the Study Visit could not be collected or participants who were considered not evaluable at the Study Visit).
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT set who were assigned to a DRC-adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 27.2 [21.2 to 33.9]

8. Secondary Outcome: Investigator Assessed Overall Response at Day 42
Description: Investigator-assessed overall response (as determined by the Investigator using all available assessment results including clinical, mycological and radiologic results based on the EORTC/MSG criteria) at Day 42, categorised by the same response criteria as in the primary endpoint: Success (Success-Complete, Success-Partial), Failure (Failure-Stable, Failure-Progression, Death, participants for whom data at Day 42 could not be collected or who were considered not evaluable at the specific visit).
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT set who were assigned to a DRC-adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 24.8 [19.0 to 31.3]

9. Secondary Outcome: Investigator Assessed Overall Response at Day 84
Description: Investigator-assessed overall response (as determined by the Investigator using all available assessment results including clinical, mycological and radiologic results based on the EORTC/MSG criteria) at Day 84, categorised by the same response criteria as in the primary endpoint: Success (Success-Complete, Success-Partial), Failure (Failure-Stable, Failure-Progression, Death, participants for whom data at Day 84 could not be collected or who were considered not evaluable at the specific visit).
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT set who were assigned to a DRC-adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 29.7 [23.5 to 36.5]

10. Secondary Outcome: DRC Adjudicated Clinical Response at Day 42
Description: DRC adjudicated clinical response at the Day 42 Study Visit, as determined by an independent Data Review Committee using clinical response results based on EORTC/MSG criteria. Resolution is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 59.9 [52.8 to 66.7]

11. Secondary Outcome: DRC Adjudicated Clinical Response at Day 84
Description: DRC adjudicated clinical response at the Day 84 Study Visit, as determined by an independent DRC using clinical response results based on EORTC/MSG criteria. Resolution is defined as a Complete or Partial Response.
Time Frame: Day 84 in the Main phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 54.0 [46.8 to 61.0]

12. Secondary Outcome: Investigator Assessed Clinical Response at Day 42
Description: Investigator assessed clinical response at the Day 42 Study Visit using clinical response results based on the EORTC/MSG criteria. Resolution is defined as a Complete or Partial Response.
Time Frame: Day 42 in the Main phase of study treatment
Population: The mITT set contains all patients in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 53.5 [46.3 to 60.5]

13. Secondary Outcome: Investigator Assessed Clinical Response at Day 84
Description: Investigator assessed clinical response at the Day 84 Study Visit using clinical response results based on the EORTC/MSG criteria. Resolution is defined as a Complete or Partial Response.
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 56.4 [49.3 to 63.4]

14. Secondary Outcome: DRC Adjudicated Mycological Response at Day 42
Description: DRC adjudicated mycological response was assessed at the Day 42 Study Visit, as determined by an independent Data Review Committee using mycological response results based on EORTC/MSG criteria. Success is defined as eradication or presumed eradication.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 18.3 [13.1 to 24.4]

15. Secondary Outcome: DRC Adjudicated Mycological Response at Day 84
Description: DRC adjudicated mycological response was assessed at the Day 84 Study Visit, as determined by an independent DRC using mycological response results based on EORTC/MSG criteria. Success is defined as eradication or presumed eradication.
Time Frame: Day 84 in the Main phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 22.5 [16.9 to 28.9]

16. Secondary Outcome: Investigator Assessed Mycological Response at Day 42
Description: Mycological response was assessed by the Investigator at the Day 42 Study Visit using mycological response results based on EORTC/MSG criteria. Success is defined as eradication or presumed eradication.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 25.7 [19.9 to 32.3]

17. Secondary Outcome: Investigator Assessed Mycological Response at Day 84
Description: Mycological response was assessed by the Investigator at the Day 84 Study Visit using mycological response results based on EORTC/MSG criteria. Success is defined as eradication or presumed eradication.
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all participants in the Intent to Treat analysis set who were assigned to a Data Review Committee adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Response rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Response rate percentage | 31.7 [25.3 to 38.6]

18. Secondary Outcome: DRC Adjudicated Radiological Response at Day 42
Description: In participants for whom radiology formed a part of their diagnosis, radiology evaluations were required on Day 42 and were adjudicated by an independent DRC. Radiological responses were assigned as per EORTC/MSG criteria.
Time Frame: Day 42 in the Main phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Count of Participants; unit: Participants
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Participants
  At least 90 percent improvement | 11
  At least 50 to less than 90 percent improvement | 10
  At least 25 to less than 50 percent improvement | 12
  Stable findings (0 to less than 25 percent improvement) | 55
  Worsening response | 6
  No signs on Radiological images at Screening | 7
  Not evaluable | 75
  Not relevant | 2
  Missing | 0
  Death (from any cause) | 24

19. Secondary Outcome: DRC Adjudicated Radiological Response at Day 84
Description: In participants for whom radiology formed a part of their diagnosis, radiology evaluations were required on Day 84 and were adjudicated by an independent DRC. Radiological responses were assigned as per EORTC/MSG criteria.
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Count of Participants; unit: Participants
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Participants
  At least 90 percent improvement | 14
  At least 50 to less than 90 percent improvement | 11
  At least 25 to less than 50 percent improvement | 5
  Stable findings (0 to less than 25 percent improvement) | 36
  Worsening response | 6
  No signs on Radiological images at Screening | 5
  Not evaluable | 71
  Not relevant | 2
  Missing | 21
  Death (from any cause) | 31

20. Secondary Outcome: Investigator Assessed Radiological Response at Day 42
Description: In participants for whom radiology formed a part of their diagnosis, radiology evaluations were required on Day 42. Radiological responses were assessed by the Investigator using EORTC/MSG criteria.
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Count of Participants; unit: Participants
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Participants
  At least 90 percent improvement | 10
  At least 50 to less than 90 percent improvement | 20
  At least 25 to less than 50 percent improvement | 20
  Stable findings (0 to less than 25 percent improvement) | 29
  Worsening response | 11
  No signs on Radiological images at Screening | 3
  Not evaluable | 69
  Missing | 16
  Death (from any cause) | 24

21. Secondary Outcome: Investigator Assessed Radiological Response at Day 84
Description: In participants for whom radiology formed a part of their diagnosis, radiology evaluations were required on Day 84. Radiological responses were assessed by the Investigator using EORTC/MSG criteria.
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all participants in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Count of Participants; unit: Participants
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Participants
  At least 90 percent improvement | 23
  At least 50 to less than 90 percent improvement | 16
  At least 25 to less than 50 percent improvement | 16
  Stable findings (0 to less than 25 percent improvement) | 26
  Worsening response | 10
  No signs on Radiological images at Screening | 4
  Not evaluable | 52
  Missing | 24
  Death (from any cause) | 31

22. Secondary Outcome: All Cause Mortality Rate at Day 42
Description: The all cause mortality rate at Day 42 uses the survival status that was entered at the study visit (which employs a window around each nominal study day).
Time Frame: Day 42 in the Main Phase of study treatment
Population: The mITT set contains all patients in the Intent to Treat analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Mortality rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Mortality rate percentage | 11.9 [7.8 to 17.2]

23. Secondary Outcome: All Cause Mortality Rate at Day 84
Description: The all cause mortality rate at Day 84 uses the survival status that was entered at the study visit (which employs a window around each nominal study day).
Time Frame: Day 84 in the Main Phase of study treatment
Population: The mITT set contains all patients in the ITT analysis set who were assigned to a DRC adjudicated disease category.
Measure: Number (95% Confidence Interval); unit: Mortality rate percentage
Arm/Group | Olorofim (F901318)
Number analyzed (Participants) | 202
Mortality rate percentage | 16.3 [11.5 to 22.2]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from the time of Informed consent through study completion, up to and including 4-week post-treatment follow-up. For patients in the main treatment phase of the study only, the median duration of study treatment was 84 days. For those entering the extended treatment phase, the median duration of study treatment was 308 days (approximately 10 months).
Description: Treatment emergent (TE) AEs occurring in main or extended phase are summarised here and defined as any AE which started or worsened on or after the first dose of main phase study treatment up to and including the post-treatment follow-up for the extended phase.
Arm/Group | Olorofim (F901318)
All-Cause Mortality (participants affected / at risk) | 50/203
Serious Adverse Events (participants affected / at risk) | 132/203
Other Adverse Events (participants affected / at risk) | 186/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olorofim (F901318) (N=203)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (2)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Acute myeloid leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Aneurysm (Vascular disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1)
Apheresis (Surgical and medical procedures) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Arthritis fungal (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
Aspergillus infection (Infections and infestations) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 2 (2)
Blastic plasmacytoid dendritic cell neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Bone marrow transplant (Surgical and medical procedures) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Candida infection (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebrospinal fluid reservoir placement (Surgical and medical procedures) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CNS ventriculitis (Infections and infestations) | 1 (1)
Coccidioidomycosis (Infections and infestations) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Complications of transplanted lung (Injury, poisoning and procedural complications) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
COVID-19 (Infections and infestations) | 8 (8)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Device breakage (Product Issues) | 1 (1)
Device leakage (Product Issues) | 1 (1)
Device malfunction (Product Issues) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Disseminated aspergillosis (Infections and infestations) | 1 (1)
Disseminated coccidioidomycosis (Infections and infestations) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Embolism (Vascular disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Exophthalmos (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Fungal endocarditis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Graft versus host disease in lung (Immune system disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hepatic enzyme increased (Investigations) | 7 (10)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Hydrocephalus (Nervous system disorders) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Liver function test increased (Investigations) | 7 (7)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Meningism (Nervous system disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Meningitis coccidioides (Infections and infestations) | 5 (6)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Mycetoma mycotic (Infections and infestations) | 1 (2)
Mycobacterium chelonae infection (Infections and infestations) | 1 (1)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Papilloedema (Eye disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Picornavirus infection (Infections and infestations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 13 (13)
Pneumonia fungal (Infections and infestations) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 2 (2)
Purulent discharge (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 9 (11)
Renal abscess (Infections and infestations) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhodococcus infection (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 4 (5)
Sepsis (Infections and infestations) | 2 (2)
Septic arthritis staphylococcal (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 4 (5)
Shunt malfunction (Injury, poisoning and procedural complications) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2)
Spinal cord compression (Nervous system disorders) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thalamic stroke (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Toxic cardiomyopathy (Cardiac disorders) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Urosepsis (Infections and infestations) | 2 (2)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Wound sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olorofim (F901318) (N=203)
Abdominal pain (Gastrointestinal disorders) | 13 (17)
Acute kidney injury (Renal and urinary disorders) | 15 (15)
Anaemia (Blood and lymphatic system disorders) | 12 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (14)
Constipation (Gastrointestinal disorders) | 15 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (19)
COVID-19 (Infections and infestations) | 18 (19)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14)
Depression (Psychiatric disorders) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 42 (51)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Fatigue (General disorders) | 18 (19)
Headache (Nervous system disorders) | 32 (42)
Hepatic enzyme increased (Investigations) | 18 (22)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (11)
Hypertension (Vascular disorders) | 11 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (13)
Hypotension (Vascular disorders) | 16 (21)
Liver function test increased (Investigations) | 22 (27)
Nausea (Gastrointestinal disorders) | 40 (53)
Oedema peripheral (General disorders) | 19 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (14)
Pyrexia (General disorders) | 29 (41)
Rash (Skin and subcutaneous tissue disorders) | 11 (13)
Urinary tract infection (Infections and infestations) | 17 (24)
Vomiting (Gastrointestinal disorders) | 40 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
F2G retains the right to review all articles referring to olorofim and generated from sponsored studies. All articles should be submitted to F2G for review at least 8 weeks prior to submission to the target journal. F2G reserves the right to delay publication or presentation if there is an issue relating to protecting intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT03583164/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03583164/SAP_001.pdf